CLINICAL TRIAL: NCT00775528
Title: An Open Label, Multi-center, Study to Assess the Safety and Tolerability of Pancrelipase Delayed Release Capsules in Infants and Children Less Than 7 Years of Age With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Brief Title: Study Investigating a Delayed-Release Pancrelipase in Patients With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Djenane Bennett, Solvay Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S245.3.128
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-10

CONDITIONS: Cystic Fibrosis; Pancreatic Exocrine Insufficiency
Keywords: Cystic Fibrosis; Pancreatic Exocrine Insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Pancrelipase Delayed Release

INTERVENTIONS:
Drug: Pancrelipase Delayed Release — 3,000, 6,000 and 12,000 unit Lipase Capsules

SUMMARY:
This study will assess the safety and tolerability of pancrelipase delayed release capsules in subjects up to 6 years of age with Pancreatic Exocrine Insufficiency (PEI) due to Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Cystic Fibrosis (CF) diagnosis by two positive chloride sweat tests or gene analysis
* Current or historical human fecal elastase < 50µg/gstool
* Weight greater than 3.75 kg
* Age 1 month to 6 years
* Currently receiving treatment with a commercially available pancreatic enzyme product on a stable dose for more than 3 months
* Clinically stable condition without evidence of acute respiratory disease or any other acute condition

Exclusion Criteria:

* Ileus or acute abdomen
* History of fibrosing colonopathy, Celiac disease, gastrectomy, Crohn´s disease and small bowel surgery other than minor resection due to meconium ileus without resulting in malabsorption syndrome
* History of distal ileal obstruction syndrome within 6 months of enrollment
* Use of an immunosuppressive drug
* Any type of malignancy involving the digestive tract in the last 5 years
* Known infection with HIV

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (12):
- United States (12):
  - Site 11, Boise, Idaho
  - Site 5, Louisville, Kentucky
  - Site 9, Boston, Massachusetts
  - Site 6, Ann Arbor, Michigan
  - Site 12, Detroit, Michigan
  - Site 4, Minneapolis, Minnesota
  - Site 13, Long Branch, New Jersey
  - Site 8, Albuquerque, New Mexico
  - Site 1, Cincinnati, Ohio
  - Site 10, Oklahoma City, Oklahoma
  - Site 7, Oklahoma City, Oklahoma
  - Site 3, Hershey, Pennsylvania

REFERENCES:
- [Background] Graff GR, McNamara J, Royall J, Caras S, Forssmann K. Safety and tolerability of a new formulation of pancrelipase delayed-release capsules (CREON) in children under seven years of age with exocrine pancreatic insufficiency due to cystic fibrosis: an open-label, multicentre, single-treatment-arm study. Clin Drug Investig. 2010;30(6):351-64. doi: 10.2165/11533390-000000000-00000. PMID 20441244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in 9 centers in US between April 2009 and June 2009. During the period of screening (Days -21 to Days -7), subjects were evaluated for eligibility. They underwent a short period of up to 7 days on their usual pancreatic enzyme supplementation before receiving the study treatment.
Pre-assignment Details: Nineteen subjects were consented and 18 subjects were allocated to pancrelipase delayed release capsule. One subject did not meet the fecal elastase requirement and did not receive study medication.
Groups:
- Pancrelipase Delayed-Release Capsules: Target dose of 8000 lipase units/kg/day. This dose was administered in divided doses with meals/snacks.
Period: Overall Study
Arm/Group | Pancrelipase Delayed-Release Capsules
Started | 19 (Started means number of patients who consented)
Completed | 18
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pancrelipase Delayed-Release Capsules
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: months] — The Baseline characteristics are presented on the Full Analysis Set meaning patients having taken the study drug and with Post-baseline efficacy data
  months | 27.3 (21.9)
Sex: Female, Male [Count of Participants; unit: Participants] — The Baseline characteristics are presented on the Full Analysis Set meaning patients having taken the study drug and with Post-baseline efficacy data
  Participants
    Female | 5
    Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Secondary Outcome: Stool Fat (% Fat)
Description: The stool fat content was calculated as percent fat of dry solid weight per bowel movement. Stool fat per patient was derived as mean over three bowel movements sampled (i.e. one sample per day).
Time Frame: Last 3 days in a 10-day treatment period
Population: The efficacy results are presented on the Full Analysis Set meaning patients having taken the study drug and with Post-baseline efficacy data.
Measure: Mean (Standard Deviation); unit: Percentage of fat
Arm/Group | Pancrelipase Delayed-Release Capsules
Number analyzed (Participants) | 18
Percentage of fat | 28.11 (9.86)

2. Secondary Outcome: Fat Intake (g)
Description: The mean daily fat intake was determined as the average of daily fat intake over a 3-day period.
Time Frame: Last 3 days in a 10-day treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Pancrelipase Delayed-Release Capsules
Number analyzed (Participants) | 18
Grams | 46.61 (22.34)

3. Secondary Outcome: Total Calorie Intake (kcal)
Description: The total calorie intake was determined as the average of total calorie of daily food intake intake over a 3-day period.
Time Frame: Last 3 days in a 10-day treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kcal
Arm/Group | Pancrelipase Delayed-Release Capsules
Number analyzed (Participants) | 18
Kcal | 1239.71 (605.78)

4. Primary Outcome: Number of Patients With at Least One Treatment Emergent Adverse Event (TEAE)
Description: Treatment Emergent Adverse Events are defined as adverse events started at or after the first administration of study drug and include those events started prior to the first administration but which worsened after the first intake.
Time Frame: 10 Days
Measure: Number; unit: Participants
Arm/Group | Pancrelipase Delayed-Release Capsules
Number analyzed (Participants) | 18
Participants | 9

ADVERSE EVENTS:
Time Frame: The adverse events presented were collected from start of drug treatment to the end of the treatment period.
Arm/Group | Pancrelipase Delayed-Release Capsules
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 9/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pancrelipase Delayed-Release Capsules (N=18)
Diarrhoea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Irritability (General disorders) | 1
Skin candida (Infections and infestations) | 1
Otitis media (Infections and infestations) | 3
Otitis media accute (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At 60 days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy and allow Sponsor 60 days to review and comment.